CLINICAL TRIAL: NCT05972356
Title: The Effect of Left Ventricular DIastolic Dysfunction on Short Term Cardiac Surgery Outcomes in Female Cardiac patieNts
Brief Title: Effect of Left Ventricle Diastolic Dysfunction on Outcomes in Female Cardiac Surgery Patients
Acronym: EDISON
Status: Not yet recruiting | Type: Observational
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Responsible Party: Principal Investigator, Jennifer Breel, drs., Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Other Study IDs: W23_003#23.024
Record Dates: First submitted 2023-07-24; First posted 2023-08-02 (Actual); Last update posted 2023-08-02 (Actual); Status verified 2023-07

CONDITIONS: Left Sided Heart Failure
Keywords: sex-differences; left ventricular diastolic dysfunction; cardiac surgery; outcomes
MeSH Terms: conditions — Heart Failure; Ventricular Dysfunction, Left

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of this study is to evaluate the differences between males and females with LVDD, undergoing cardiac surgery. We will look at perioperative factors such as body weight, body surface area, previous medical history, cardiac function measured by amongst others, transoesophageal echocardiography and haemodynamic parameters, transfusion, coagulation, cardiopulmonary bypass (CPB) related factors, inotropic requirements, risk, and outcome scores as well as complications, morbidity and mortality at 30 days. We will evaluate these variables in an observational setting, with the goal of improving outcome in females after cardiac surgery in the future.

DETAILED DESCRIPTION:
Cardiovascular disease is the leading cause of death among females in the Netherlands. According to the Netherlands Heart Registry (NHR), 25% more females than males died as a result of cardiovascular disease in 2019. In addition, females who undergo a cardiac surgery intervention have a higher risk of morbidity and mortality after cardiac surgery than males.1

An important predictor and risk factor of adverse outcomes after cardiac surgery is the perioperative presence of heart failure (HF) with preserved ejection fraction (EF) (HFpEF).

HFpEF, also known as left ventricular diastolic dysfunction (LVDD), accounts for 30-50% of all patients presenting with symptoms of HF.2 Two-thirds of these patients are female.3 The incidence of LVDD is generally increases with age.4 However, females are more likely to develop LVDD than males of the same age (ratio 2:1).5 Vascular stiffening is a crucial pathophysiological factor that contributes to the higher prevalence of LVDD in females. Females show a faster decline of ventricular elastance with age compared with males.6 Furthermore, several comorbidities contribute to a higher prevalence of LVDD in females: iron deficiency, diabetes, obesity, hypertension, preeclampsia, and autoimmune diseases. All are associated with the onset of an inflammatory response, which is considered as an important factor in the development of LVDD.6

In diagnosing LVDD and determining its severity, echocardiography is of crucial value. Indeed, echocardiographic imaging allows LVDD to be classified into grades ranging from grade I (mild) to grade III (severe). In this regard, a higher grade is equivalent to a higher likelihood of symptomatic HF, and a worse prognosis. Transoesophageal echocardiography is the standard-of-care perioperative diagnostic intervention during cardiac surgery operations, to assess cardiac function. Intraoperatively, the simplified algorithm of Swaminathan et al.,8 is used to assess diastolic function.

Several studies investigated sex-related differences in the outcomes of patients with LVDD, who were treated conservatively. 9-12 These studies demonstrated that females with LVDD had similar outcomes of in-hospital and all-cause mortality compared with males. However, none of these studies focused on outcomes after cardiac surgery.

Additionally - despite known differences leading to higher morbidity and mortality in females after cardiac surgery - basic and clinical research has predominantly included male animals and male patients.

The aim of this study is to evaluate the differences between males and females with LVDD, undergoing cardiac surgery. We will look at perioperative factors such as body weight, body surface area, previous medical history, cardiac function measured by amongst others, transoesophageal echocardiography and haemodynamic parameters, transfusion, coagulation, cardiopulmonary bypass (CPB) related factors, inotropic requirements, risk, and outcome scores as well as complications, morbidity and mortality at 30 days. We will evaluate these variables in an observational setting, with the goal of improving outcome in females after cardiac surgery in the future.

We hypothesise that LVDD is more pronounced in female patients compared to male patients. Additionally, we hypothesise that females with LVDD (dependent on the grade of LVDD) have a poorer early outcome (≤30 days) after cardiac surgery than male patients.

ELIGIBILITY:
Inclusion Criteria:

* All patients >18 years, who undergo cardiac surgery from 1 January 2023 till 31 December 2026 in the Amsterdam UMC

Exclusion Criteria:

* Patients who object to the re-use of their care data

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients undergoing cardiac surgery will be asked for permission to use data collected as standard-of-care
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2023-07-25 (Estimated); Primary Completion 2026-07-25 (Estimated); Study Completion 2027-07-25 (Estimated)

PRIMARY OUTCOMES:
Left ventricular diastolic dysfunction | Before statrt bypass and end of bypass
  number of patients with LVDD (grade I - III) before and after CPB. LVDD is measured by using the ratio of trans-mitral early flow velocity to early mitral annular tissue velocity (E/E')

SECONDARY OUTCOMES:
Composite endpoint | measured 30 days after surgery
  Composite endpoint: Mortality,Cerebrovascular accident (CVA), with persistent neurological disability, Acute kidney injury (AKI), as defined by KDIGO 2012,Low cardiac output syndrome (LCOS) with a vasoactive-inotropic score (VIS) > 45 or need for cardiac assist device,Pulmonary (and other) complications requiring ventilation >48 hours

CONTACTS AND LOCATIONS:
Overall Officials: Markus W Hollmann, Prof.Dr.Dr., Principal Investigator — Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)

IPD SHARING:
Plan to Share IPD: Undecided